CLINICAL TRIAL: NCT04999202
Title: An Open-label, Phase 1b, Dose Escalation and Expansion Study to Evaluate the Safety, Tolerability, Maximum Tolerated or Administered Dose, Pharmacokinetics, Pharmacodynamics and Efficacy of the Aryl Hydrocarbon Receptor Inhibitor (AhRi) BAY 2416964 in Combination With Pembrolizumab in Participants With Advanced Solid Tumors
Brief Title: A Study to Learn How Safe the Study Drug BAY 2416964 (AhR Inhibitor) in Combination With the Treatment Pembrolizumab is, How This Combination Affects the Body, the Maximum Amount That Can be Given, How it Moves Into, Through and Out of the Body and Its Action Against Advanced Solid Cancers in Adults
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Last patient ongoing on treatment ended the study on 20th January 2025. Hence, the end of study was reached as defined in the protocol.
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 21343; PN-A61 (Other: Merck); 2023-503547-33-00 (Other: CTIS (EU)); 2020-003547-28 (EudraCT Number)
Record Dates: First submitted 2021-08-05; First posted 2021-08-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Advanced Solid Tumors
Keywords: Non-small cell lung cancer (NSCLC); Head and neck squamous cell carcinoma (HNSCC); Urothelial Cancer; Advanced cancer; Immunotherapy; Immuno oncology; Aryl Hydrocarbon Receptor inhibitor(AhRi); Aryl Hydrocarbon Receptor; Pembrolizumab; aPD1; Checkpoint inhibitor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose escalation of BAY2416964 (Experimental): Six dose levels of BAY 2416964 (as determined in the first in human mono-therapy study of BAY2416964) are planned in combination with standard dose Pembrolizumab.
  Interventions: Drug: BAY2416964; Drug: Pembrolizumab
- Dose expansion of BAY2416964 in tumor type specific cohort (Experimental): To determine the RP2D of BAY2416964 in combination therapy with pembrolizumab. Participants will be enrolled in up to 3 tumor type-specific cohorts including relapsed/refractory non-small cell lung cancer (NSCLC), head and neck squamous cell carcinoma (HNSCC) and urothelial cancer.
  Interventions: Drug: BAY2416964; Drug: Pembrolizumab

INTERVENTIONS:
Drug: BAY2416964 — Oral, twice or three times daily
  Arms: Dose escalation of BAY2416964
Drug: BAY2416964 — The highest dose determined safe in combination with pembrolizumab in the dose escalation part or a lower dose. More than one dose may be explored in the dose expansion.
  Arms: Dose expansion of BAY2416964 in tumor type specific cohort
Drug: Pembrolizumab — Administered as a dose of 200 mg using a 30-minute IV infusion every 3 weeks

SUMMARY:
Researchers are looking for a better way to treat advanced solid cancers including head and neck cancer, lung cancer and bladder cancer.

In some people with cancer a protein called Aryl Hydrocarbon Receptor (AhR) can prevent immune cells from fighting tumor cells. The study drug, BAY 2416964, is a small molecule which blocks the AhR allowing the body to use its immune response against the cancer cells. Researchers think that BAY 2416964 given together with a cancer treatment called pembrolizumab may help shrink tumors in people with cancer.

The main aims of this study are to find for BAY 2416964 in combination with pembrolizumab,

* how safe this drug combination is
* how it affects the body (also referred to as tolerability)
* the highest amount of BAY 2416964 that can be given in combination with pembrolizumab without too many side effects.

The researchers will also study the action of BAY 2416964 in combination with pembrolizumab against the cancer.

The participants in this study will get BAY 2416964 and pembrolizumab. BAY 2416964 will be given by mouth. Pembrolizumab will be given as an intravenous (IV) infusion. An IV infusion is given through a needle into a vein.

This study will have two parts. The first part will help find the most appropriate dose that can be given in the second part.

Each participant of the first, so called dose escalation part, will be assigned to one specific dose group for BAY 2416964. The amount of BAY 2416964 that is given changes step-wise from one group to the next. The dose of pembrolizumab will always be the same.

The participants of the second, so called dose expansion part, will receive the most appropriate dose of BAY 2416964 found in the first part.

During the study, the participants will receive the treatment in 3-week periods called cycles. In each cycle, the participants will in general get pembrolizumab once and BAY 2416964 in a daily schedule. These 3-week cycles will be repeated throughout the trial. The participants can take the study treatment until their cancer gets worse, until they have medical problems, or until they leave the trial. Participants will have around 4 visits in each cycle. Some of the visits can also be done via phone.

During the study, the study doctors and their team will:

* take blood and urine samples
* check if the participants' cancer has changed in size using computed tomography scans or magnetic resonance imaging scans of the participants' tumors
* check the participants' overall health
* ask the participants questions about how they are feeling and what adverse events they are having.

An adverse event is any medical problem that a participant has during a study. Doctors keep track of all adverse events that happen in studies, even if they do not think the adverse events might be related to the study treatments.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥18 years of age inclusive, at the time of signing the informed consent.
* Participants with following histologically or cytologically confirmed advanced solid tumors that have progressed after treatment with all available therapies for metastatic disease that are known to confer clinically meaningful benefit, or are intolerant to treatment, or refuse standard treatment.

  * Dose Escalation: all solid tumor types
  * Tumor type-specific Expansion cohorts:

    * NSCLC
    * HNSCC with primary location in oropharynx, oral cavity, hypopharynx or larynx
    * Urothelial Cancer
* Participants must have progressed on treatment with an anti-PD-1/L1 monoclonal antibody (mAb) administered either as monotherapy, or in combination with other checkpoint inhibitors or other therapies.
* Have measurable disease per RECIST 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.

Exclusion Criteria:

* Severe (Common terminology criteria for adverse events (CTCAE) v.5 Grade ≥ 3) infections within 4 weeks before the first study intervention administration
* Active autoimmune disease that has required systemic treatment in past 2 years
* Has a diagnosis of immunodeficiency or is receiving immunosuppressive therapy
* Has active Central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Cardiac disease as specified in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
The incidence of TEAEs including TESAEs | After first administration of BAY2416964 in combination with pembrolizumab up to 90 days after the last dose of BAY2416964 in combination with pembrolizumab
  TEAEs: treatment-emergent adverse events TESAEs: treatment-emergent serious adverse events
The severity of TEAEs including TESAEs | After first administration of BAY2416964 in combination with pembrolizumab up to 90 days after the last dose of BAY2416964 in combination with pembrolizumab
Maximum tolerated dose (MTD) or maximum administered dose (MAD) of BAY2416964 | Cycle 1 (21 days) in dose escalation
  The MTD/MAD is the dose level that can be safely given, defined as the occurrence of dose-limiting toxicities (DLTs) below a certain threshold.

SECONDARY OUTCOMES:
Cmax of BAY2416964 after single-dose in Cycle 1 | Cycle 1 Day 1 (1 cycle is 21 days)
Cmax of BAY2416964 after multiple-dose in Cycle 1 | Cycle 1 Day 15 (1 cycle is 21 days)
AUC(0-t) (t depend on the dosing regimen) of BAY2416964 after single-dose in Cycle 1 | Cycle 1 Day 1 (1 cycle is 21 days)
AUC(0-t) (t depend on the dosing regimen) of BAY2416964 after multiple-dose in Cycle 1 | Cycle 1 Day 15 (1 cycle is 21 days)
Objective response rate (ORR) by Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1) | At the end of Cycle 2 (-7 days, each cycle is 21 days), Cycle 4 (-7 days) and at the end of every third cycle (-7 days) from Cycle 5 onwards
  ORR will be evaluated using RECIST 1.1 by investigator assessment.

CONTACTS AND LOCATIONS:
Locations (14):
- United States (6):
  - Florida Cancer Specialists, Altamonte Springs, Florida
  - Florida Cancer Specialists & Research Institute, Sarasota, Florida
  - Brigette Harris Cancer Pavilion at Henry Ford Cancer Center - Detroit, Detroit, Michigan
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology- Austin Midtown, Austin, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
- Italy (5):
  - IRCCS Istituto Nazionale Tumori Fondazione Pascale - S. C. Sperimentazioni Cliniche, Napoli, Campania
  - Fondazione IRCCS Istituto Nazionale dei Tumori - S. C. Oncologia Medica 1, Milan, Lombardy
  - Istituto Europeo di Oncologia s.r.l - Sviluppo di nuovi farmaci per Terapie Innovative, Milan, Lombardy
  - ASST Grande Ospedale Metropolitano Niguarda, Milan, Lombardy
  - Humanitas Mirasole S.p.A. - Oncologia Medica ed Ematologia, Rozzano, Lombardy
- National University Hospital Medical Centre, Singapore, Singapore
- United Kingdom (2):
  - Belfast City Hospital, Belfast, North Ireland
  - Freeman Hospital, Newcastle, Tyne and Wear

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.